CLINICAL TRIAL: NCT03469596
Title: Evaluation by MRI of Anal Canal Cell Carcinoma: is There Predictive Factor?
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: IRMcanalANAL
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Anal Carcinoma
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI sequence — several MRI sequence before and after contrast product injection.

SUMMARY:
Anal canal cell carcinoma is a very rare cancer but well treated. If the morphological test are well established in the initial evaluation, it's not the case of the follow up evaluation particularly by MRI.About 1/3 of patient decline with metastatic relapse during the follow up of these patients.It appears that clinical regression seen precociously is a predictive factor of survival without relapse. But there 's no study confirming that point.

This context takes us to evaluate if there is a predictive factor in MRI to final clinical result.

ELIGIBILITY:
Inclusion Criteria:

* patient with anal canal cell carcinoma histologically proved
* patient with initial MRI and follow up MRI in Hospital St Joseph's radiology yard.
* patient for whom a radio chemotherapy treatment decision was taken.

Exclusion Criteria:

* patients with already metastatic lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient with anal canal cell carcinoma with an initial MRI in GHPS between 1st august 2009 and 24th april of 2015
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Distance with regard to the anal margin | maximum of 6 years after the initial MRI
  tumor position
initial tumor size | maximum of 6 years after the initial MRI
  Maximal tumoral size in the cranio-caudal plan in cm
presence of nodal status | maximum of 6 years after the initial MRI
  presence of nodal status in inguinal region

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France